CLINICAL TRIAL: NCT03234933
Title: Post-Operative Ambulatory Challenge and Exercise (PACE) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael T. Jaklitsch, Michael Jaklitsch, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-152
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobility Tracker (Experimental): * Each patient will be provided by the research team staff with a new mobility tracker
  * The standard pre-operative assessment, surgical procedure and post-operative care will still be done
  * Measurements of each patient (steps, distance and calories) will be obtained by the research staff
  Interventions: Other: Mobility Tracker

INTERVENTIONS:
Other: Mobility Tracker — Tracking Patient's movements and calories

SUMMARY:
This research study is evaluating the postoperative results in terms of quality of life and functional recovery of elderly patients after cancer surgery.

DETAILED DESCRIPTION:
This is a pilot study, designed to collect data on steps walked (ambulation) per day of lobectomy patients after surgery. While the investigators know ambulation improves outcomes after surgery, there is no institutional policy, set of patient goals, or method for deciding which patients require further resources, such as physical therapy. Data collected will be used to set up a hospital-wide strategy for patients to achieve post-operative ambulation milestones more readily.

ELIGIBILITY:
Inclusion Criteria:

* Patients Aged ≥ 18 years
* Who underwent or who will undergo lung resection at Brigham and Women's Hospital (BWH)
* With diagnosis of malignant or benign disease

Exclusion Criteria:

* Patients with baseline immobility (i.e. wheelchair-bound, use of any walking assistance device, or gait alterations)
* Patients with cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Steps Taken | 2 years
  Number of steps taken by subjects will be recorded on a mobility tracker, starting at the time of admission to the floor and ending at the time of discharge.

SECONDARY OUTCOMES:
Distance walked | 2 years
  The distance walked by subjects will be recorded on a mobility tracker, starting at the time of admission to the floor and ending at the time of discharge.
Number of Calories Burned | 2 years
  The number of calories burned by subjects will be recorded on a mobility tracker, starting at the time of admission to the floor and ending at the time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Jaklitsch, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No